CLINICAL TRIAL: NCT04966416
Title: The Effect of Orally Administered Pyrophosphate on Calcinosis Formation in Systematic Sclerosis
Brief Title: Calcinosis Reduction by Pyrophosphate in SSC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Szeged University (Other)
Collaborators: Research Centre for Natural Sciences (Other); University of Debrecen Dept. of Rheumatology (Unknown)
Responsible Party: Principal Investigator, László Kovács MD, PhD, Professor, Szeged University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CALC-001
Record Dates: First submitted 2021-07-14; First posted 2021-07-19 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Systemic Sclerosis; Scleroderma
Keywords: calcinosis; pyrophosphate
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse; Calcinosis | interventions — diphosphoric acid

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pyrophosphate (Experimental): Disodium pyrophosphate
  Interventions: Dietary Supplement: Pyrophosphate
- Placebo (Placebo Comparator): Glucose
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Pyrophosphate — 50 mg/kg bwt once daily in gelatine capsules.
  Arms: Pyrophosphate
Dietary Supplement: Placebo — Glucose in gelatine capsules.
  Arms: Placebo

SUMMARY:
Calcinosis, i.e. crystal-like nodules are troublesome complication of systemic sclerosis, an autoimmune disease. Pyrophosphate inhibits its formation is laborytory. We would like to test if orally administered pyrophosphate prevents calcinosis formation.

DETAILED DESCRIPTION:
Calcinosis, the formation of hydroxyapatite subcutaneous nodules, often complicates systemic sclerosis. There is no standard treatment for it. Based upon our preclinical experienc, we would like to test it orally administered pyrophosphate inhibits calciosis.

ELIGIBILITY:
Inclusion Criteria:

* to meet ACR/ EULAR classification criteria

Exclusion Criteria:

* severe upper minfestation of SSC
* hypo- or hyperthyreoidism
* QT prolongation on ECG

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in the size of calcinosis nodues. | 52 weeks+ 16 weeks
  Volumetric assessment with low energy CT

SECONDARY OUTCOMES:
Change of the severity of sympthoms caused by calcinosis | 52 weeks+ 16 weeks
  Visual analogue scale (0-100)
Change of the activity of calcinosis | 52 weeks+ 16 weeks
  Visual analogue scale (0-100)
Change of the size of calcinosis by ultrasound | 52 weeks+ 16 weeks
  Volumetric assessment by ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: László Kovács, MD, Ph.D., Principal Investigator — Szeged University; András Váradi, PhD, DSc, Study Director — Department of Enzymology, Research Centre for Natural Sciences

REFERENCES:
- [Background] Hsu VM, Kozak E, Li Q, Bocskai M, Schlesinger N, Rosenthal A, McClure ST, Kovacs L, Balint L, Szamosi S, Szucs G, Carns M, Aren K, Goldberg I, Varadi A, Varga J. Inorganic pyrophosphate is reduced in patients with systemic sclerosis. Rheumatology (Oxford). 2022 Mar 2;61(3):1158-1165. doi: 10.1093/rheumatology/keab508. PMID 34152415
- [Background] Dedinszki D, Szeri F, Kozak E, Pomozi V, Tokesi N, Mezei TR, Merczel K, Letavernier E, Tang E, Le Saux O, Aranyi T, van de Wetering K, Varadi A. Oral administration of pyrophosphate inhibits connective tissue calcification. EMBO Mol Med. 2017 Nov;9(11):1463-1470. doi: 10.15252/emmm.201707532. PMID 28701330